CLINICAL TRIAL: NCT03151356
Title: Value of Prostate Health Index for Prostate Cancer Diagnosis
Brief Title: Prostate Health Index for Prostate Cancer Diagnosis
Acronym: PHI-1
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0203
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients addressed for prostate biopsies because of clinical and/or biological suspicion of prostate cancer.
  Interventions: Device: Measurement of Prostate Health Index (PHI)

INTERVENTIONS:
Device: Measurement of Prostate Health Index (PHI) — Use of a diagnostic tool to predict prostate biopsy outcome: measurement of total and free PSA as well as the [-2]proPSA and calculation of The Prostate Health Index according to the following formula: Prostate Health Index (PHI) = [p2PSA /fPSA] x √tPSA

SUMMARY:
Prostate biopsies are the gold standard for prostate cancer (PCa) diagnosis. They are performed according to the results of the measurement of prostate-specific antigen (PSA) in the serum of patients with PCa suspicion. More than half of the prostate biopsies reveal eventually negative because of the poor specificity of prostate-specific antigen assay. The Prostate Health Index (PHI) is a new diagnostic tool that has been described as a good predictor of prostate biopsy outcome. No large study has been performed so far in France. This study aim to evaluate Prostate Health Index diagnostic performances in a large multicentric French cohort of patients undergoing prostate biopsies because of clinical and/or biological suspicion of prostate cancer.

Prostate Health Index will be measured in patients directed to prostate biopsies according to usual practices. Inclusion of 400 patients within 6 months in 12 French centers is expected. The ability of Prostate Health Index to predict prostate cancer at biopsy will be evaluated in terms of intrinsic and extrinsic diagnostic performances including sensitivity, specificity, predictive values, diagnostic accuracy, area under receiver operating curves and decision curve analyses.

ELIGIBILITY:
Inclusion Criteria:

* Man ≥ 18 years old
* Addressed for prostate biopsy because of serum total Prostate Specific Antigen ≥ 4 ng/mL and/or abnormal digital rectal examination and/or first degree familial history of prostate cancer
* Agreeing to participate to the study

Exclusion Criteria:

* Personal history of positive prostate biopsy (evidence of prostate cancer)
* Personal history or evidence of prostate cancer based on clinical data (highly suspicious digital rectal examination (≥cT3) and/or serum total PSA ≥ 20 ng/mL and/or evidence for lymph node or bone metastases (retroperitoneal lymph nodes, bone lesions …)
* Evidence for synchronous non-prostate cancer (current active treatment)
* Adult protected by law

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients addressed for prostate biopsies because of prostate cancer suspicion: serum total Prostate Specific Antigen ≥ 4 ng/mL and/or abnormal digital rectal examination and/or first degree familial history of prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Intrinsic performances of Prostate Health Index in predicting prostate biopsy outcome | When the results of all prostate biopsies will be available (approximately at 7 months after the beginning of the study)
  Area under receiver operating curve (ROC) analysis; the ROC curve will be constructed from the values of the sensitivity and specificity of Prostate Health Index by comparison to the gold standard, i.e. prostate biopsy outcome (cancer or not).

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Mondor, Créteil
  - CHU Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Clinique Louvière de Lille, Lille
  - Hôpital Edouard Herriot, Lyon
  - Clinique Beau Soleil, Montpellier
  - Hôpital Tenon, Paris
  - Unité Médicale d'Oncologie et de Transfert - Service de Biochimie et Biologie Moléculaire - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - CHU de Rennes, Rennes
  - Clinique Atlantis, Saint-Herblain
  - IUCT Oncopole de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No